CLINICAL TRIAL: NCT02166125
Title: Endoscopic Sutures For Gastrointestinal Tract Disorders: A Prospective Multicenter Registry.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief of Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1207012584
Record Dates: First submitted 2014-06-10; First posted 2014-06-18 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Endoscopic Suturing Within the Gastrointestinal Tract
Keywords: gastric bypass; sleeve gastrectomy; esophageal stent; suturing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic suturing: Any patient who has undergone clinically indicated and/or standard of care endoscopic suturing within the Gastrointestinal tract.
  Interventions: Procedure: Endosuturing

INTERVENTIONS:
Procedure: Endosuturing — Endoscopic suturing

SUMMARY:
The purpose of this prospective registry is to assess long term data on efficacy, safety and clinical outcome of endoscopic placement of suture(s) and approximation of soft tissue within the Gastrointestinal tract for various GI tract disorders. The registry will evaluate technical feasibility, clinical outcome, safety profile and overall clinical management through medical chart review. The procedures the investigators are evaluating are all clinically indicated and will not be prescribed to someone to participate in this research study.

DETAILED DESCRIPTION:
Our institution performs therapeutic Interventional Endoscopy in around 500-1000 patients a year. We come across several gastrointestinal disorders such as fistula or leak repairs, gastric outlet revisions, (dilated anastomoses), stent migrations, gastric wall defects or perforation, ulcer repairs, closure of transgastric entrance after a NOTES procedure (Natural orifice translumenal endoscopic surgery) that require placement of sutures and/or approximation of soft tissue.

Conventionally, surgery or other endoscopic alternatives are used to resolve or mitigate these issues. However, surgery had higher morbidity and mortality rates, and other endoscopic alternatives may not be successful either.

With the advent of endoscopic suture systems such as the Apollo Endosurgery OverStitch™ Endoscopic Suture System (ESS) (or Endo Stitch™ , the SILS™ Stitch), advanced endoscopists can place endoscopic sutures by deploying multiple running and interrupted stitches with a single insertion of the endoscope within the gastrointestinal tract.

Currently, the endoscopy unit uses the Apollo Endosurgery OverStitch™ Endoscopic Suture System (ESS) for suture placement in various gastrointestinal disorders; including suturing stents to prevent stent migration in the esophagus. Even though several case reports and animal studies have been published reporting the clinical success of endoscopic suturing, there have been hardly any large sample size studies to verify the safety and efficacy of endoscopic suturing. Our own study reported 12 cases with promising results for esophageal stent subjects. 1-16 We lack enough data evaluate and verify technical feasibility, clinical success and safety of endoscopic suturing in specific gastrointestinal disorders.1-16 Evaluation of these factors would help us compare them to conventional treatment modalities; and consequently help us identify appropriate treatment techniques and improve clinical management of patients.

The purpose of this prospective registry is to assess long term data on efficacy, safety and clinical outcome of endoscopic placement of suture(s) and approximation of soft tissue within the Gastrointestinal tract for various GI tract disorders. The registry will evaluate technical feasibility, clinical outcome, safety profile and overall clinical management through medical chart review. The procedures we are evaluating are all clinically indicated and will not be prescribed to someone to participate in this research study.

Study Design: Prospective, observational, medical chart review for at least 6 standard of care visits up to 1 year after subject consents for study participation.

Interventions: None

Subject Participation: Subject's participation in this study will allow us to collect data for at least 6 standard of care visits up to 1 year after consenting to participating in this registry study.

Subject will undergo a standard of care or clinically indicated Endoscopic procedure and subsequent follow up clinic visits as part of their standard medical care. Subject will sign a separate clinical consent for the Endoscopic procedure and placement of the sutures(s). That consent form will explain the procedure as well as the risks involved with the procedure.

Subject will undergo endoscopic suturing and subsequent follow up clinic visits regardless of their participation in this study. Subject will undergo no additional tests and procedures as part of this study.

This registry study allows for the prospective review and collection of clinical data related to endoscopic suturing for safety and efficacy assessment.

Study duration: At least 6 standard of care visits up to 1 year for each subject

* Once the subject consents, data will be collected for their clinically indicated or standard of care procedure visit and follow up visits.
* Standard of care follow up visits for endoscopic suturing are usually 1 month, 3 months and 6 months post procedure. No additional research related visits will be requested.
* All data will be collected from Medical charts.
* No subject surveys or questionnaires will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone clinically indicated and/or standard of care endoscopic suturing within the Gastrointestinal tract
* Above or equal to 18 years of age

Exclusion Criteria:

* Any patient who has not undergone endoscopic suturing within the gastrointestinal tract
* Below 18 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who has undergone clinically indicated and/or standard of care endoscopic suturing within the Gastrointestinal tract.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-05-26 (Estimated); Study Completion 2017-08-26 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 6 months to 1 year
  Documentation of technical success and clinical outcome rates. Technical success will be documented via number of sutures successfully placed. Clinical success will be documented via follow up of resolution of symptoms of primary indication and number of repeat interventions or other interventions for the same indication.

SECONDARY OUTCOMES:
Safety Outcome | 30 days post procedure
  Documentation of Safety: Number of Participants with Adverse Events; Type, frequency and intensity of adverse events.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ochsner Health Center - Kenner, Kenner, Louisiana
  - Weill Cornell Medical College, New York, New York
  - Digestive Health Associates of Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
No IPD sharing